**Study Title:** User Evaluation of the Guide To Goals Application - a Care Coordination Tool to Translate ADA Clinical Standards of Care for Children with T2D into Practice

**Document Title:** Minor Assent Form (version 2)

**NCT:** NCT03926598

Document Approval Date: 04/01/2020

# ASSENT DOCUMENT FOR ENROLLING MINORS IN A RESEARCH STUDY

Georgia Institute of Technology
Project Title: User Evaluation of the Guide-To-Goals
Application - a Care Coordination Tool to Translate ADA
Clinical Standards of Care for Children with T2D into
Practice

Investigators: Dr. Jiten Chhabra MD, MS

You are being asked to be in a research study. Your mom/parent/guardian knows about the study, but you can decide if you want to be in it or not.

## **Purpose:**

- We are trying to understand whether an Ipad app developed by Georgia Tech researchers for patients, families and caregivers of children with Type 2 Diabetes called Guide-To-Goals is easy to use or not.
- Results from this work will help researchers make this application easier to use.
- You may guit at any time during the study if you want to.
- We expect to include 10 people in the study.

## What Will Be Done:

- If you decide to be in this study, your mom/parent/guardian will bring you to the Children's Healthcare of Atlanta Diabetes Clinic once. Your mom/parent/guardian will be here in the room with you the whole time.
- First we will let you try our app on our Ipad for 15 minutes and ask you to do certain tasks on the app like logging in and selecting or unselecting check boxes within the app. During this time we will see you use the app and take notes.
- After that we will ask you a few questions about your experience using the app and help you fill out a questionnaire with 5 simple questions.
- The entire session will not last more than 1 hour.

### **Risks/Discomforts:**

We don't think you will be uncomfortable or hurt at all
while being in this study. If you want to stop using the app
or not answer our questions, that's OK and nobody will be
angry or disappointed.

# **Benefits:**

• We don't think that being in this study will help you at all with your Type 2 Diabetes. We hope to learn how to help other children with Type 2 Diabetes by making easy to use apps.

# To Thank You:

• There will be no compensation for participants, but we thank all participants for their contributions and time.

#### **Confidentiality:**

• We won't tell your friends or teachers or anyone besides your mom/parent/guardian that you are in this study.

## In Case of Injury/Harm:

• If you get hurt as a result of being in this study, your mom/parent/guardian has been told what to do.

# Participant Rights:

- You don't have to be in this study if you don't want to be.
- You can stop being in the study any time.
- Nobody will be angry or disappointed if you decide not to be in the study or if you decide to quit.

### **Questions:**

• You can ask Dr. Jiten Chhabra anything about the study by calling 404-630-3787. You can also call the Georgia Tech Office of Research Integrity Assurance at 404 / 894-6942 or 404 / 385-2175 if you have questions.

| If you want to be in the study, please sign on the line below.<br>Remember, you can quit being in the study any time. | |
|---|---|
| Participant Name (printed) | _ |
| Participant Signature | Date |
| Signature of Person Obtaining Consent | Date |